CLINICAL TRIAL: NCT00992667
Title: Inhaled Apocynin Decreases Reactive Oxygen Species Concentrations in Exhaled Breath Condensate in Mild Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Rafal Pawliczak, Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nowak-01
Record Dates: First submitted 2009-10-05; First posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Bronchial Asthma
Keywords: apocynin; asthma
MeSH Terms: conditions — Asthma | interventions — acetovanillone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthmatics (Experimental): Ten nonsmoking patients, suffering from mild bronchial asthma participated in the study (mean age 30±9 years, 5 men, 5 women). Asthma was diagnosed based on GINA 2008 criteria. The patients were free of any medication, at least 7 days before, and had not suffered from any infectious diseases including upper respiratory tract infections for at least 3 months prior to the study. Patients who did not meet these criteria were excluded from the study.
  Interventions: Drug: Apocynin nebulization

INTERVENTIONS:
Drug: Apocynin nebulization — 6 ml of apocynin of total dose 3 mg (0.5 mg/ml dissolved in sterile 0.9% NaCl as the study drug) has been nebulized for 15-20 min through the mouthpiece with using of a nose clip. A nebulizer Pulmo Aide AP-50 (DeVilbiss; Richmond, VA) was used (mass median aerosol diameter 3.1 mm, output 0.3 ml/min.)
  Other Names: 4-hydroxy-3-methoxyacetophenone,; acetovanillone

SUMMARY:
The aim of the study is to investigate the effect of inhaled apocynin on ROS (reactive oxygen species) and NOS (reactive nitrogen species) synthesis in 10 nonsmoking mild asthmatics. Effects of nebulized apocynin (0.5 mg/ml, 6 ml) are assessed in exhaled breath condensate (EBC) after 30, 60 and 120 minutes.

DETAILED DESCRIPTION:
The study had a double-blind, placebo-controlled, cross-over design, consisted of 2 visits, separated 30 ± 10 days. If during the first visit the drug was used, in the second visit - placebo or vice versa. Before and after procedure, safety measures (arterial blood pressure, heart rate value, and cough scale) were performed. The effect of a possible inhibitor of ROS formation was performed using corticosteroid-naive asthmatic subjects, which are more prone to oxidative stress than healthy non-smoking subjects. The study protocol was approved by the Ethics Committee of Medical University of Lodz (no. RNN/12/08/KE) and written consent was obtained from every subject prior to the study.

EBC was collected using a modification of the method described previously by Doniec et al.2005. The subjects breathed spontaneously through a mouthpiece for 20 min. Each subject wore a nose clip during this procedure. Approximately 2 ml of condensate was collected and immediately stored at -80°C until the procedure of H2O2, NO2- and NO3- measurement.

6 ml of apocynin of total dose 3 mg (0.5 mg/ml) has been nebulized through the mouthpiece with using of a nose clip.

The H2O2 concentration in EBC was measured according to the method applied previously by Nowak et al.2001. Determination of NO2- and NO3- with Griess solution was performed by micromethod, carried out in 96-well plates, according to Griess' method, modified the method described by Dziedzic et al.2003.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from bronchial asthma (mild)
* patients free of any medication at least 7 days before research
* patients had not suffered from any infectious diseases including upper respiratory tract infections for at least 3 months prior to the study

Exclusion Criteria:

* patients suffering from moderate or severe asthma
* patients taking medication 7 or less days before the study
* infectious diseases that had occurred 3 months or less before the study

Ages: 22 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
blood pressure, peripheral blood differential count, lung functional tests, single breath carbon monoxide diffusing capacity | 6 months

SECONDARY OUTCOMES:
determination of H2O2, NO2- and NO3- concentrations in exhaled breath condensate, determination of NO2 concentration in serum, blood pressure, peripheral blood differential count, lung functional tests, single breath carbon monoxide diffusing capacity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Pawliczak, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

REFERENCES:
- [Background] Horvath I, Hunt J, Barnes PJ, Alving K, Antczak A, Baraldi E, Becher G, van Beurden WJ, Corradi M, Dekhuijzen R, Dweik RA, Dwyer T, Effros R, Erzurum S, Gaston B, Gessner C, Greening A, Ho LP, Hohlfeld J, Jobsis Q, Laskowski D, Loukides S, Marlin D, Montuschi P, Olin AC, Redington AE, Reinhold P, van Rensen EL, Rubinstein I, Silkoff P, Toren K, Vass G, Vogelberg C, Wirtz H; ATS/ERS Task Force on Exhaled Breath Condensate. Exhaled breath condensate: methodological recommendations and unresolved questions. Eur Respir J. 2005 Sep;26(3):523-48. doi: 10.1183/09031936.05.00029705. PMID 16135737
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595
- [Background] Dziedzic B, Mazanowska-Gajdowicz J, Walczewska A, Sarniak A, Nowak D. Comparison of cadmium and enzyme-catalyzed nitrate reduction for determination of NO2-/NO3- in breath condensate. Clin Chim Acta. 2003 Sep;335(1-2):65-74. doi: 10.1016/s0009-8981(03)00277-8. PMID 12927686
- [Result] Peters EA, Hiltermann JT, Stolk J. Effect of apocynin on ozone-induced airway hyperresponsiveness to methacholine in asthmatics. Free Radic Biol Med. 2001 Dec 1;31(11):1442-7. doi: 10.1016/s0891-5849(01)00725-0. PMID 11728816
- [Result] Nowak D, Kalucka S, Bialasiewicz P, Krol M. Exhalation of H2O2 and thiobarbituric acid reactive substances (TBARs) by healthy subjects. Free Radic Biol Med. 2001 Jan 15;30(2):178-86. doi: 10.1016/s0891-5849(00)00457-3. PMID 11163535
- [Derived] Gage MC, Thippeswamy T. Inhibitors of Src Family Kinases, Inducible Nitric Oxide Synthase, and NADPH Oxidase as Potential CNS Drug Targets for Neurological Diseases. CNS Drugs. 2021 Jan;35(1):1-20. doi: 10.1007/s40263-020-00787-5. Epub 2021 Jan 30. PMID 33515429